CLINICAL TRIAL: NCT01227083
Title: Comparison of the Responsiveness of Two Different Asthma-specific QOL Measures (AQLQ and cAQOL) in Korean Patients With Persistent Asthma
Brief Title: 2nd_Computerized Asthma Specific Quality of Life(cAQOL)
Acronym: 2nd_cAQOL
Status: Completed | Type: Observational
Sponsor: Ajou University School of Medicine (Other)
Collaborators: Yonsei University (Other); Inha University Hospital (Other); Dong-A University (Other)
Responsible Party: Principal Investigator, Hae-Sim Park, Professor, Department of Surgery, Ajou University School of Medicine, Ajou University School of Medicine
Other Study IDs: AJIRB-GEN-OBS-10-178
Record Dates: First submitted 2010-10-22; First posted 2010-10-25 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Persistent Asthma Patient
Keywords: AQLQ and cAQOL

STUDY DESIGN:
Biospecimen Retention: Samples With DNA — Sub-group of ADRB2 and NK2R genotypes
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Asthma control test check AQLQ(Asthma Quality of Life Questionnaire)after being cAQOL(Computerized Asthma specific quality of life)
- 2: Asthma control test check cAQOL(Computerized Asthma specific quality of life)after being AQLQ(Asthma Quality of Life Questionnaire)

SUMMARY:
Comparison of the responsiveness of two different asthma-specific QOL measures (AQLQ and cAQOL) in Korean patients with persistent asthma

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 20-70 years
* Patient diagnosed with asthma over six months ago
* Asthma diagnosis

  * Airway reversibility, FEV1 ≥ 12% and 200mL or
  * Airway hyper-responsiveness, PC20 < 16 mg/mL or
  * More than two weeks, more than 2 times a day in excess of 20% PEFR diurnal variability patient
* FEV1 55-100% of predicted value patient
* Inhaled corticosteroids alone or inhaled corticosteroids and beta agonists used patient
* Currently, at least if you have one or more asthma symptoms, asthma control test (ACT • Asthma Control Test) score of less than 19 characters
* Patients who sufficiently listen to the purpose and content of this trial and the properties of investigational products and voluntarily agree with the participation to sign a written consent approved by IRB of Ajou University Medical Center before the participation in this trial

Exclusion Criteria:

* Current smoking or smoking in the past 15packyears
* Patients who show a symptom of an acute disease within 14 days before the beginning of this trial (administration of trial medication)
* Recent changes in asthma treatment for 28days
* Chronic diseases that affect the quality of life

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: asthma control patient
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2010-10; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Two asthma quality of life measurement tool | 24 weeks treatment
  Two asthma quality of life measurement tool (cAQOL, AQLQ) and the correlation between ACT

SECONDARY OUTCOMES:
Correlation between cAQOL/AQLQ | treatment screening, week1,week12,week24
  -Correlation between cAQOL/AQLQ and other clinical parameters including FEV1, and asthma exacerbation.
Association of asthma control therapy and a questionnaire | 24 weeks treatment
  -The proportion of subjects with achieving well controlled asthma within ACT & cAQOL-guided management strategy with ICS or ICS/LABA based on GINA 2006 guidelines during 24 weeks.
asthma patient genotypes | Screening
  Sub-group of ADRB2 and NK2R genotypes

CONTACTS AND LOCATIONS:
Overall Officials: Hae-Sim Park, MD,PhD, Principal Investigator — Ajou University School of Medicine
Locations (1):
- Ajou University Medical Center, Suwon, South Korea